CLINICAL TRIAL: NCT06772428
Title: A Prospective, Randomized, Parallel-controlled Clinical Study of Nano-crystalline Megestrol Acetate Combined With Standard Treatment Versus Standard Treatment Alone for Adjuvant Therapy in Patients With High-risk Factor Squamous Cell Carcinoma of the Head and Neck After Surgery.
Brief Title: Nano-crystalline Megestrol Acetate for Adjuvant Treatment in High-risk Head and Neck Squamous Cell Carcinoma After Surgery.
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Changchun GeneScience Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Megaxia ES-HNSCC-01
Record Dates: First submitted 2024-12-25; First posted 2025-01-13 (Actual); Last update posted 2025-01-13 (Actual); Status verified 2024-12

CONDITIONS: Head and Neck Squamous Cell Carcinoma; Underwent Surgery Within 6 Weeks and Postoperative Assessment Indicated High-risk Factors

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Nano-crystalline Megestrol Acetate Oral Suspension + Standard Therapy (Experimental)
  Interventions: Drug: Nano-crystalline Megestrol Acetate Oral Suspension; Radiation: standard treatment
- Standard Therapy (Active Comparator)
  Interventions: Radiation: standard treatment

INTERVENTIONS:
Drug: Nano-crystalline Megestrol Acetate Oral Suspension — Nano-crystalline Megestrol Acetate Oral Suspension, with a specification of 125 mg/mL, the study group takes 5 mL orally per day (625 mg/day), and continues medication; after completing the treatment cycle, patients who are assessed by the researchers as suitable for continued treatment may continue to receive therapy.
  Arms: Nano-crystalline Megestrol Acetate Oral Suspension + Standard Therapy
Radiation: standard treatment — radiotherapy ± chemotherapy

SUMMARY:
This study is a prospective, randomized, parallel-controlled clinical trial, with the primary objective to evaluate the efficacy and safety of nano-crystalline megestrol acetate combined with standard treatment compared to standard treatment alone for adjuvant therapy in patients with high-risk squamous cell carcinoma of the head and neck (excluding nasopharyngeal carcinoma) after surgery.

ELIGIBILITY:
Inclusion Criteria:

* ≥18 years at the time of enrollment.
* Eastern Cooperative Oncology Group (ECOG) performance status score of 0-2.
* Life expectancy ≥6 months.
* Patients with histologically or cytologically confirmed squamous cell carcinoma of the head and neck (oral cavity, oropharynx, larynx, and hypopharynx).
* Patients who have undergone surgery for head and neck squamous cell carcinoma within 6 weeks and are assessed postoperatively as having high-risk factors requiring radiotherapy ± chemotherapy.

Exclusion Criteria:

* Suffering from tumors in areas other than the oral cavity, oropharynx, larynx, and hypopharynx, such as nasopharyngeal carcinoma or other unknown primary head and neck tumors.
* Having any condition that affects gastrointestinal absorption, such as dysphagia, malabsorption, or uncontrollable vomiting; currently undergoing tube feeding or parenteral nutrition.
* Suffering from anorexia due to neurosis, mental illness, or difficulty eating due to pain.
* Suffering from Acquired Immune Deficiency Syndrome (AIDS).

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 96 (Estimated)
Dates: Start 2025-01-01 (Estimated); Primary Completion 2027-06-30 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
The proportion of subjects with improved appetite based on A/CS-12 assessment | Week 3
The proportion of subjects with a relative increase in body weight of >5% from baseline | Week 12

CONTACTS AND LOCATIONS:
Locations (1):
- West China School of Medicine/West China Hospital of Sichuan University, Chengdu, Sichuan, China